CLINICAL TRIAL: NCT00758342
Title: A Double-Masked, Parallel-Group, Efficacy and Safety Study of Brinzolamide 1.0% (AZOPT) as Adjunctive Therapy to Travoprost 0.004% (TRAVATAN) in Patients With Chronic Angle-Closure Glaucoma
Brief Title: Azopt (Brinzolamide 1.0%) Plus Travatan (Travoprost 0.004%) in Treating Patients With Chronic Angle-Closure Glaucoma (CACG)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty of enrolling patients
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-06-01
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2010-02-05 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2010-02

CONDITIONS: Intraocular Pressure
Keywords: IOP lowering efficacy and safety of Azopt plus Travatan
MeSH Terms: interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travoprost 0.004% + Brinzolamide 1.0% (Experimental): Travoprost 0.004% (once daily) + Brinzolamide 1.0% (twice daily)
  Interventions: Drug: Travoprost 0.004% + Brinzolamide 1.0%
- Travoprost 0.004% + Tears Natural (Active Comparator): Travoprost 0.004% (once daily) + Tears Naturale (twice daily)
  Interventions: Drug: Travoprost 0.004% + Tears Natural

INTERVENTIONS:
Drug: Travoprost 0.004% + Brinzolamide 1.0% — Travoprost 0.004% (once daily) + Brinzolamide 1.0% (twice daily)
  Arms: Travoprost 0.004% + Brinzolamide 1.0%
Drug: Travoprost 0.004% + Tears Natural — Travoprost 0.004% (once daily) + Tears Naturale (twice daily)
  Arms: Travoprost 0.004% + Tears Natural

SUMMARY:
To evaluate the IOP (Intraocular Pressure) lowering efficacy and safety of Brinzolamide 1.0% (Azopt), dosed twice daily as adjunctive therapy in patients treated with Travoprost 0.004% (Travatan) once daily. The study is double masked. The patients will receive either treatment for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years;
* CACG (Chronic Angle Closure Glaucoma) ≥ 1eye
* have been treated with PGA (prostaglandin analogues) once daily ≥ 2 weeks prior to the screening visit and IOP=19-32 mmHg (millimeters mercury) in at least one eye and ≤ 32 mmHg in both eyes
* clinical stability of VA (Visual Acuity) and optic nerve throughout the study

Exclusion Criteria:

* Abnormality restricts exam of the fundus or anderior chamber
* conjunctivitis, keratitis or uveitis
* unable to be discontinued from using all ocular hypotensive medication(s) except Travatan (Travoprost 0.004%) and/or Azopt (Brinzolamide 1.0%) for 12days-4weeks
* ocular surgery prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Travoprost 0.004% + Brinzolamide 1.0%: Travoprost 0.004% + Brinzolamide 1.0%
- Travoprost 0.004% + Tears Natural: Travoprost 0.004% + Tears Natural
Period: Overall Study
Arm/Group | Travoprost 0.004% + Brinzolamide 1.0% | Travoprost 0.004% + Tears Natural
Started | 19 | 18
Completed | 15 | 17
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travoprost 0.004% + Brinzolamide 1.0% | Travoprost 0.004% + Tears Natural | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 15 | 26
  >=65 years | 8 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean IOP (Intraocular Pressure)
Time Frame: Screening: Week 12; (At 9 am and 4 pm time points)
Measure: Mean (Standard Deviation); unit: mm Hg (millimeters mercury)
Arm/Group | Travoprost 0.004% + Brinzolamide 1.0% | Travoprost 0.004% + Tears Natural
Number analyzed (Participants) | 19 | 18
mm Hg (millimeters mercury)
  9 AM measurement | 17.58 (4.29) | 20.59 (3.70)
  4 PM measurement | 17.11 (4.50) | 18.50 (3.05)

ADVERSE EVENTS:
Arm/Group | Travoprost 0.004% + Brinzolamide 1.0% | Travoprost 0.004% + Tears Natural
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: Other
Confidentiality agreement